CLINICAL TRIAL: NCT02129894
Title: The Use of Abdominal Binders in Patients Undergoing Cesarean Sections: A Randomized Controlled Trial
Brief Title: The Use of Abdominal Binders in Patients Undergoing Cesarean Sections
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLHN-50-14
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Cesarean Section Post Operative Management
Keywords: cesarean section; postoperative pain; pregnancy; abdominal binder
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- abdominal binder (Active Comparator): Post cesarean section patients will get a abdominal binder placed
  Interventions: Device: abdominal Binder
- No Abdominal Binder (No Intervention): Post cesarean section patients will not have abdominal binder

INTERVENTIONS:
Device: abdominal Binder — placement of abdominal binder
  Arms: abdominal binder

SUMMARY:
To see if the use of Abdominal Binders improves patients out comes after cesarean delivery

DETAILED DESCRIPTION:
Inclusion: All patients admitted to labor and delivery

Consented patients who had a cesarean delivery will be randomized using a number table to receive or not receive an abdominal binder.

Outcomes: On postoperative days 1 and 2, patients were asked to complete a pain visual analog scale and the validated Symptom Distress Scale. Postoperative hemoglobin and hematocrit were also recorded.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing cesarean section for any indication

Exclusion Criteria:

* unable to give consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Pain measurement | up to post operateive day 2
  Pain will be measured using a visual analog scale
Patient Distress score | up to post operateive day 2
  A validated patient distress score will be used

SECONDARY OUTCOMES:
hemoglobin and hematocrit | post operative day 1 and 2
Pain medication usage | post operative day 1 and 2

CONTACTS AND LOCATIONS:
Locations (1):
- St Luke's University Hospital, Bethlehem, Pennsylvania, United States

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021
- [Derived] Gillier CM, Sparks JR, Kriner R, Anasti JN. A randomized controlled trial of abdominal binders for the management of postoperative pain and distress after cesarean delivery. Int J Gynaecol Obstet. 2016 May;133(2):188-91. doi: 10.1016/j.ijgo.2015.08.026. Epub 2016 Jan 14. PMID 26892694